CLINICAL TRIAL: NCT07194226
Title: Attitudes and Decision Regret Regarding Fertility Preservation in Transgender Individuals
Acronym: Fertilitrans
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Maria Cristina Meriggiola, Prof., IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: Fertilitrans_v1
Record Dates: First submitted 2025-08-29; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-07

CONDITIONS: Fertility Preservation in Transgender Persons
Keywords: Fertility preservation; Decision regret; Transgender adults; Gender-affirming treatment
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational survey; participants complete an anonymous questionnaire and no medical or behavioral intervention is applied.

SUMMARY:
The goal of this observational survey is to learn how transgender adults think and feel about saving their fertility before gender-affirming treatment. We will ask at least 300 participants in Emilia-Romagna to answer an anonymous online questionnaire. The main questions are:

* Why did people choose or decline fertility preservation?
* How much regret do they feel about their decision?
* What counseling or support did they receive, and was it helpful?
* What personal or financial factors influenced their choice?

This study will help doctors and counselors improve fertility-preservation advice for transgender adults in Italy.

DETAILED DESCRIPTION:
Background & Rationale

For transgender individuals, fertility is particularly complex because gender-affirming treatments such as hormone therapy, hysterectomy, or orchiectomy can permanently impact reproductive potential. At our center, fertility preservation through gamete (egg or sperm) or gonadal tissue cryopreservation is routinely offered before initiating these treatments.

However, no studies in Italy have explored why transgender individuals choose to preserve or not preserve fertility, nor how satisfied or regretful they feel about these choices afterward. Understanding the motivations, barriers, and emotional outcomes around these decisions is crucial to providing truly informed, person-centered counseling that respects transgender individuals' reproductive autonomy and supports their overall quality of life.

This study aims to fill this gap by exploring these critical aspects within the Italian transgender community to improve fertility-preservation counseling practices.

Study Objectives & Hypotheses

Primary Objective: Measure decision regret (5-item Decision Regret Scale) and identify factors-such as counseling quality and life changes-that predict higher regret.

Hypothesis: Higher regret scores will be found in those declining preservation or receiving less comprehensive counseling.

Secondary Objectives:

* Characterize primary motivations (e.g., cost, family support) behind preservation decisions.
* Describe counseling experiences by modality (in-person vs. telehealth), provider type, and satisfaction.
* Document barriers (medical, financial, logistical, dysphoria-related) encountered during preservation or use of gametes.
* Assess participants' preferences and attitudes toward future fertility-preservation counseling and procedures.

Methods & Questionnaire

This cross-sectional, observational survey will enroll ≥600 transgender adults (≥18 years) via:

* Clinical Recruitment: routine care patients at the Unit of Gynecology and Human Reproduction Pathophysiology, IRCCS AOU Bologna
* Community Recruitment: anonymous REDCap questionnaire distributed in UNIBO departmental atria and through regional social-media outlets

The questionnaire covers:

* Demographics & Transition History (age, sex assigned at birth, gender identity, education, employment, hormone/surgery timeline)
* Fertility-Preservation Decision
* For those who preserved: procedure type, timing, encountered difficulties, satisfaction, and non-use reasons.
* For those who did not: main reasons and attitudes toward future preservation.
* Counseling Experience: modality, provider role, and satisfaction rating.
* Decision Regret Scale (DRS, 5-item): validated measure of post-decision regret.
* Psychosocial Context: relationship status, social support, economic situation, and life satisfaction.

Statistical Analysis Plan Primary Outcome (DRS): compute mean, SD, and distribution; compare by preservation status (t-test) and counseling quality (ANOVA); multivariate linear regression adjusting for age, support, and other covariates.

Secondary Outcomes:

* Motivations: report proportions; analyze associations with regret (chi-square, logistic regression).
* Counseling Satisfaction: summarize frequencies; correlate with DRS.
* Barriers: tabulate reported obstacles; test relationships with psychological impact (chi-square).
* Preferences & Attitudes: describe proportions and conduct subgroup comparisons.

Additional Analyses: sensitivity checks for missing data (imputation), interaction/subgroup analyses (e.g., changes in relationship or finances).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as transgender
* Age ≥ 18 years.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified transgender individuals of any sex assigned at birth, at any stage of gender affirmation
Study Population: The study population consists of adult transgender individuals followed in routine clinical practice at the Unit of Gynecology and Human Reproduction Pathophysiology, IRCCS AOU Bologna, and the general transgender population of the Emilia-Romagna region reached via questionnaire distribution in the atria of UNIBO departmental buildings and through social-media networks.
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Decision Regret Scale (DRS) Score (5-Item) | Through study completion, approximately three months.
  Scores collected with the 5-item Decision Regret Scale to assess participants' levels of regret about their fertility-preservation choice. Includes analysis of regret frequency by type and quality of counseling received and identification of personal factors (e.g., marital status, social support) that may have contributed to regret.

SECONDARY OUTCOMES:
Frequency of Main Motivations for Fertility Preservation Decision | Through study completion, approximately three months.
  Frequency of the primary reasons (e.g., cost, family support, personal priorities) for choosing or declining fertility preservation and their association with Decision Regret Scale scores.
Counseling Modalities and Satisfaction | Through study completion, approximately three months.
  Distribution of counseling types received (modality and provider) and participants' satisfaction ratings regarding the adequacy and helpfulness of fertility-preservation counseling.
Barriers to Fertility Preservation and Psychological Impact | Through study completion, approximately three months.
  Percentage and types of difficulties reported during gamete preservation and use.
Preferences and Attitudes Toward Counseling and Fertility Preservation | Through study completion, approximately three months.
  Participants' expressed preferences and attitudes regarding counselling on fertility-preservation options.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request.